CLINICAL TRIAL: NCT06802692
Title: Determination of the Effects of Virtual Reality Glasses and Meditation Music on Anxiety, Pain, Vital Signs, Satisfaction and Pregnancy Outcomes During Embryo Transfer Procedure: a Randomized Controlled Experimental Study
Brief Title: Effects of Virtual Reality Glasses and Meditation Music on Anxiety, Pain, Vital Signs, Satisfaction and Pregnancy Outcomes in Embryo Transfer Procedure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, DİDEM KAYA, Assistant Professor, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NuhNaciYazganUdk; Nuh Naci Yazgan University (Other: Nuh Naci Yazgan University)
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Being Diagnosed with Primary Infertility; Having Had an Embryo Transfer for the First Time
Keywords: Embryo Transfer; Virtual Reality Glasses; Meditation Music; Anxiety; Pain; Vital Signs; Satisfaction; Pregnancy
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Visual reality glasses and meditation music group (Experimental): Starting 15 minutes before the ET procedure, participants in the VR glasses and meditation music group will be shown a video of the sea, underwater and forest with VR glasses and will be made to listen to meditation music. At the same time, meditation music will be played. When the ET procedure is completed, the video and meditation music will be stopped. After the procedure, the VR glasses will be disinfected with antiseptic spray before being used on another patient, and disposable ear pads will be placed on the headphones after each patient. Anxiety, pain, vital signs (pulse, diastolic blood pressure, systolic blood pressure, respiration and peripheral oxygen saturation) will be evaluated 15 minutes before and immediately after the ET procedure. 15 minutes after the ET procedure, satisfaction with the ET procedure, the application of VR glasses and listening to meditation music will be evaluated.
  Interventions: Behavioral: VR glasses and meditation music group
- Meditation music group (Experimental): Meditation music group participants will listen to meditation music through headphones starting from 15 minutes before the ET procedure until the procedure is completed. When the ET procedure is completed, the meditation music will be stopped. After the procedure, disposable ear pads will be placed on the headphones for each patient. Anxiety, pain, vital signs (pulse, diastolic blood pressure, systolic blood pressure, respiration and peripheral oxygen saturation) will be assessed 15 minutes before and immediately after the ET procedure. 15 minutes after the ET procedure, satisfaction with the ET procedure and listening to meditation music will be assessed.
  Interventions: Behavioral: Meditation music group
- Control group (No Intervention): Control group participants will not receive any intervention other than the ET procedure. Anxiety, pain, vital signs (pulse, diastolic blood pressure, systolic blood pressure, respiration, and peripheral oxygen saturation) will be assessed 15 minutes before and immediately after the ET procedure.

INTERVENTIONS:
Behavioral: VR glasses and meditation music group — Starting 15 minutes before the ET procedure, participants in the VR glasses and meditation music group will be shown a video of the sea, underwater and forest with VR glasses and will be made to listen to meditation music. At the same time, meditation music will be played. When the ET procedure is completed, the video and meditation music will be stopped. After the procedure, the VR glasses will be disinfected with antiseptic spray before being used on another patient, and disposable ear pads will be placed on the headphones after each patient. Anxiety, pain, vital signs (pulse, diastolic blood pressure, systolic blood pressure, respiration and peripheral oxygen saturation) will be evaluated 15 minutes before and immediately after the ET procedure. 15 minutes after the ET procedure, satisfaction with the ET procedure, the application of VR glasses and listening to meditation music will be evaluated.
  Arms: Visual reality glasses and meditation music group
Behavioral: Meditation music group — Meditation music group participants will listen to meditation music through headphones starting from 15 minutes before the ET procedure until the procedure is completed. When the ET procedure is completed, the meditation music will be stopped. After the procedure, disposable ear pads will be placed on the headphones for each patient. Anxiety, pain, vital signs (pulse, diastolic blood pressure, systolic blood pressure, respiration and peripheral oxygen saturation) will be assessed 15 minutes before and immediately after the ET procedure. 15 minutes after the ET procedure, satisfaction with the ET procedure and listening to meditation music will be assessed.
  Arms: Meditation music group

SUMMARY:
The aim of this study is to determine the effects of virtual reality glasses (VRG) and meditation music on anxiety, pain, vital signs, satisfaction and pregnancy outcomes during the embryo transfer (ET) procedure.

H1: VR glasses + meditation music (1st intervention group), meditation music (2nd intervention group) application has an effect on anxiety.

H2: VR glasses + meditation music (1st intervention group), meditation music (2nd intervention group) application has an effect on pain.

H3: VR glasses + meditation music (1st intervention group), meditation music (2nd intervention group) application has an effect on vital signs (pulse rate, blood pressure, respiration).

H4: VR glasses + meditation music (1st intervention group), meditation music (2nd intervention group) application has an effect on patient satisfaction.

H5: VR glasses + meditation music (1st intervention group), meditation music (2nd intervention group) application has an effect on pregnancy outcomes.

35 women will be included in the VRG+meditation group, 35 women in the meditation group, and 35 women in the control group. The first group will be shown a nature view with VRG and will listen to meditation music 15 minutes before the ET. The second group will be shown meditation music 15 minutes before the embryo transfer. No intervention will be made in the third group. In the first two groups, anxiety, pain, vital signs (pulse, diastolic blood pressure, systolic blood pressure, respiration, and peripheral oxygen saturation) will be assessed 15 minutes before and immediately after the ET procedure. In the first group, satisfaction with the ET procedure, VRG application, and listening to meditation music will be assessed 15 minutes after the ET procedure. In the second group, satisfaction with the ET procedure and listening to meditation music will be assessed 15 minutes after the ET procedure.

DETAILED DESCRIPTION:
Infertility is considered not only financially costly and psychologically stressful, but also emotionally and physically painful due to the uncertainty of diagnostic and treatment procedures as well as pregnancy outcomes (Kızılkaya et al. 2024). In vitro fertilization (IVF-ET) with embryo transfer is an effective treatment for infertility worldwide (Gu et al 2019). Embryo transfer (ET), being the final and critical step of the IVF cycle, can often cause anxiety and pain in couples (Federica Di Guardo & Marco Palumbo 2022; Saravelos et al. 2016). Women are likely to experience anxiety and depression at the end of long and uncertain treatment processes (Federica Di Guardo & Marco Palumbo 2022). The patient's bladder should be full before the ET procedure. This can help both to visualize the uterus more clearly on ultrasound and to facilitate the passage of the transfer catheter by correcting the anteverted uterus. However, patients complain of significant discomfort and pain due to their full bladder, especially when the ultrasound probe is pressed against the abdomen (Frishman et al 2007). Pain can also be caused by passing the catheter through the cervix (Karavani et al. 2017).

Women seek information and treatment about complementary health approaches to increase their chances of conceiving, having a live birth, improving their health, quality of life, and reducing anxiety during treatment (Smith et al. 2019). In recent years, the use of complementary and alternative medicine has increased significantly because it is cost-effective, easy to access, and individuals do not have to worry about invasive procedures or side effects of chemical drugs. Virtual reality (VR) headset is defined as a computer-generated three-dimensional space in which the user is immersed. Its purpose is to provide users with the perception of being in a non-physical world and to create a sense of immersion by using head-mounted displays (HMDs) that surround them with images, sounds, or other stimuli. Intuitively, VR helps relieve symptoms of pain, stress, anxiety, and depression in an imaginary space and enables patients to achieve positive and pleasant emotions (Federica Di Guardo & Marco Palumbo 2022).

Listening to relaxing music before a stressful event affects the endocrine, autonomic, cognitive and emotional systems differently, and music-based interventions have low economic costs (Kızılkaya et al. 2024). Since music increases serotonin secretion, it makes people feel positive, reduces patient stress, increases comfort and helps them cope better with pain (Kızılkaya et al. 2024; Karaman Özlü et al. 2022). The benefits of music therapy include distracting, reducing anxiety and worry, providing pain control, reducing stress, facilitating communication, relaxing and eliminating insomnia, regulating vital signs, reducing sweating, relaxing muscles, providing easy breathing and strengthening the immune system (Karaman Özlü et al. 2022). Recent studies focusing on the relationship between psychological symptoms and pregnancy rates during Assisted Reproductive Technologies cycles have shown controversial results. Some authors have reported that the higher the stress level experienced by women before and during treatment, the lower the pregnancy rate (Klonoff-Cohen et al. 2001; An et al. 2013, Terzioğlu et al. 2016; Xu et al. 2017), while other studies have not supported the same results (Boivin et al. 2011; Pasch et al. 2012). Up to now, virtual reality and music listening applications have been used in different fields to determine pain, anxiety, vital signs and satisfaction, as well as in the field of women's health. However, very few studies have been found to reduce pain and anxiety experienced during the ET procedure. This study is the first randomized controlled trial known in the literature to investigate the effects of VR and meditation music, which are distraction methods during the embryo transfer procedure, on the anxiety, pain, vital signs, patient satisfaction and pregnancy outcomes of infertile women.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with primary infertility
* Having had an embryo transfer for the first time

Exclusion Criteria:

* Using antidepressants or sedatives
* Using painkillers within 24 hours before the procedure
* Having hearing and vision impairment

Termination Criteria:

* Removing glasses during the procedure
* Removing headphones during the procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | To be administered to women 15 minutes before the ET procedure and immediately after the ET procedure is completed (the ET procedure is 20 minutes). Change in baseline State-Trait Anxiety Scale scores at the end of 35 minutes.
  Anxiety will be assessed using the State-Trait Anxiety Scale. The original name of the scale is State-Anxiety Invertory. The scale was developed by Spielberger [1970] and adapted to Turkish by Oner and Le Compte (1983). It consists of 20 items rated on a four-point Likert-type scale. The scale describes how people feel under different conditions and at that moment. The inventory is in the form of a four-point Likert scale. The total score varies between 20 and 80, and higher scores indicate higher anxiety levels. The Cronbach's alpha value of the scale is 0.94 [1983].
VAS-Pain | Applied to women immediately before the ET procedure and immediately after the ET procedure is completed (ET procedure is 20 minutes). Change in baseline VAS-Pain scores after 20 minutes.
  Pain will be assessed using the Visual Analog Scale (VAS). The VAS is a 10 cm long horizontal line. The women marks the point on the line that they think represents their perception of their current condition. The VAS score is determined by measuring in millimeters from the left end of the line to the point marked by the women. The left most end of the line includes the expressions "no pain (0 points)" and the right most end includes the expressions "unbearable pain (10 points)" (Wewers and Lowe 1990).
Change from Baseline Pulse Rates | Pulse will be measured 15 minutes before the ET procedure and on the same day immediately after the ET procedure is completed (ET procedure is 20 minutes). Change from baseline pulse rates after 35 minutes.
  Women's pulses will be measured and recorded 15 minutes before the ET procedure and immediately after the ET procedure is completed.
Change from Baseline Blood Pressure | Blood pressure will be measured 15 minutes before the ET procedure and on the same day immediately after the ET procedure is completed (ET procedure is 20 minutes). Change from baseline blood pressure after 35 minutes.
  Women's blood pressure will be measured and recorded 15 minutes before the ET procedure and immediately after the ET procedure is completed.
Change from Baseline Respiratory Rates | Respiratory rates will be measured 15 minutes before the ET procedure and on the same day immediately after the ET procedure is completed (ET procedure is 20 minutes). Change from respiratory rates after 35 minutes.
  Women's respiratory rates will be measured and recorded 15 minutes before the ET procedure and immediately after the ET procedure is completed.
Change from Baseline Oxygen Saturation (SpO2) | Oxygen saturation will be measured 15 minutes before the ET procedure and on the same day immediately after the ET procedure is completed (ET procedure is 20 minutes). Change from oxygen saturation after 35 minutes.
  Women's oxygen saturation will be measured and recorded 15 minutes before the ET procedure and immediately after the ET procedure is completed.
VRG+meditation music group satisfaction form | This form must be filled out on the same day, 15 minutes after the ET process is completed.
  This form was prepared to determine satisfaction with the ET procedure, the video watched with the virtual reality glasses, and the meditation music listened to. The first question of the 1st intervention group asks whether they are satisfied with the virtual reality glasses application. The second question asks whether they are satisfied with the meditation music. The third question asks whether they are satisfied with the ET procedure. In these questions, women will be asked to indicate their satisfaction levels on a 10-centimeter horizontal line. The line starts with 0 (Not satisfied at all) and ends with 10 (Very satisfied). The fourth question asks whether they would like to use the virtual reality glasses if the procedure is repeated, and the fifth question asks whether they would like to listen to meditation music if the procedure is repeated. The fourth and fifth questions are answered as yes, no, and undecided.
Meditation music group satisfaction form | This form must be filled out on the same day, 15 minutes after the ET process is completed.
  This form was prepared to determine satisfaction with the ET procedure and the meditation music listened to.The first question of the 2nd intervention group asks whether they are satisfied with the meditation music. The second question asks whether they are satisfied with the ET procedure. In these questions, women will be asked to indicate their satisfaction levels on a 10-centimeter horizontal line. The line has a value of 0 (I am not satisfied at all) at the beginning and 10 (I am very satisfied) at the end. The third question asks whether they would like to listen to meditation music if the procedure is repeated. This question is answered with yes, no and undecided.
Control group ET process satisfaction form | This form must be filled out on the same day, 15 minutes after the ET process is completed.
  The control group is only asked whether they are satisfied with the ET procedure. In this question, women are asked to indicate their satisfaction levels on a 10-centimeter horizontal line. The line has a value of 0 (I am not satisfied at all) at the beginning and 10 (I am very satisfied) at the end.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] • Smith AC, Armour M, Shewamene Z, Tan HY, Norman RJ, Johnson NP (2019) Acupuncture performed around the time of embryo transfer: a systematic review and meta-analysis. RBMO; 38(3): 364-379. https://doi.org/10.1016/j.rbmo.2018.12.038 • Kızılkaya M, Karaahmet AY, Beydag KD (2024) The Effect of Music Interventions on Anxiety, Pain, and Pregnancy Rates in Women with Infertility Before Oocyte Collection and Embryo Transfer: Systematic Review and Meta analysis of Randomized Controlled Trials. European Journal of Integrative Medicine. 72. 102408. https://doi.org/10.1016/j.eujim.2024.10240 • Gu YE, Zhang X, Zhang Q, Dai MC, Wu Y, Zhou Y, Qu F (2019) The effects of acupuncture on pregnancy outcomes of in vitro fertilization with embryo transfer: An interdisciplinary systematic review. Journal of Gynecology Obstetrics Human Reproduction 48(8): 677-684. https://doi.org/10.1016/j.jogoh.2019.07.008 • Karaman Özlü Z, Yetiş Demir Z, Özlü İ, Kılınç T, Yayla A (2022) Cerrahi Hastalarında Müzik Terapinin Semptom Yönetimine Etkisi. Karya Journal Of Health Scıence. 3(3): 354-358. https://doi.org/10.52831/kjhs.1110926 • Federica Di Guardo & Marco Palumbo (2022) Immersive virtual reality as tool to reduce anxiety during embryo transfer. Journal of Obstetrics and Gynaecology. 42(5): 802-808, https://doi.org/10.1080/01443615.2021.1995855 • Saravelos SH, Wong AWY, Kong GWS, Huang J, Klitzman R, Li TC (2016) Pain duringembryotransfer isindependently associated with clinical pregnancy in fresh/frozen assisted reproductive technology cycles. The Journal of Obstetrics and Gynaecology Research, 42(6): 684-693. https://doi.org/10.1111/jog.12962 • Wewers M, Lowe N. A critical review of visual analogue scales in the measurement of clinical phenomena Research in nursing & health 1990;13:227-36. https://doi.org/10.1002/nur.4770130405 • Spielberger CD, Gorsuch RL and Lushene RE (1970) STAI Manual for the State-Trait Anxiety Inventory. Consulting Psychologists Press. • Oner N, Le Compte A. Duru
- See also: Related Info — https://doi.org/10.1016/j.rbmo.2018.12.038
- See also: Related Info — https://doi.org/10.1016/j.jogoh.2019.07.008
- See also: Related Info — https://doi.org/10.52831/kjhs.1110926
- See also: Related Info — https://doi.org/10.1016/j.fertnstert.2017.01.023
- See also: Related Info — https://doi.org/10.1016/s0015-0282(01)02008-8